CLINICAL TRIAL: NCT00182286
Title: The Evaluation of the Continuity of Care at the Group Health Centre, A Unique Multi-Specialty, Multi-Disciplinary Health Service Organization
Brief Title: Evaluation of Continuity of Care at a Health Service Organization
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Health Services Research Foundation (Other); Group Health Centre, Sault Ste Marie, ON (Unknown); Group Health Centre (Other); Ontario Ministry of Health and Long Term Care (Other Government)
Organization: McMaster University (Other)
Other Study IDs: RC 1030106
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Continuity of Care; Patient Perspective; Health Service Organization
MeSH Terms: conditions — Diabetes Mellitus | interventions — Costs and Cost Analysis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: Assessment of continuity of care from the patient perspective
Behavioral: Relationship between continuity of care, patient outcomes, and costs

SUMMARY:
This project was conducted with patients at a multi-disciplinary, multi-specialty health services organization serving 44,000 rostered patients in Northern Ontario. It investigated continuity of care for patients with diabetes in the areas of barriers and potential solutions to, and correlates of continuity; and variability in costs associated with continuity of care and patient outcomes.

DETAILED DESCRIPTION:
Continuity of care is a concept that has been garnering increased attention in the last few years. There have been multiple methods proposed by researchers for measuring continuity of care, most of which are based on proportions or ratios of visits to the same health care provider or centre. While a consistent method for measuring continuity of care is lacking, increased continuity of care using various definitions and measurement tools has been related to better well being, lower health care costs, better glucose control, and higher satisfaction but has also not been found to improve health outcomes in other scenarios. Whether a patient is better served by high sequential access to one provider or any provider within the same system or management team is controversial. Finally, patients' perceptions of continuity of care have not been generally evaluated or correlated with current measurement methods. This project was conducted with patients at the Group Health Centre in Sault Ste Marie, Ontario, a multi-disciplinary, multi-specialty health services organization serving 44,000 rostered patients

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Diagnosis of diabetes mellitus (according to the definition used in 1999 by the Canadian Diabetes Association

Exclusion Criteria:

* Gestational diabetes
* Could not communicate in English
* Life expectancy or residency expectancy in Sault Ste Marie of less than three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342
Dates: Start 1999-09; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Overall Officials: Hui Lee, MD FRCPC MSc, Principal Investigator — Group Health Centre
Locations (1):
- Group Health Centre, Sault Ste. Marie, Ontario, Canada

REFERENCES:
- [Result] Dolovich LR, Nair KM, Ciliska DK, Lee HN, Birch S, Gafni A, Hunt DL. The Diabetes Continuity of Care Scale: the development and initial evaluation of a questionnaire that measures continuity of care from the patient perspective. Health Soc Care Community. 2004 Nov;12(6):475-87. doi: 10.1111/j.1365-2524.2004.00517.x. PMID 15717895
- [Result] Nair KM, Dolovich LR, Ciliska DK, Lee HN. The perception of continuity of care from the perspective of patients with diabetes. Fam Med. 2005 Feb;37(2):118-24. PMID 15690252
- See also: Group Health Centre Website — http://www.ghc.on.ca